CLINICAL TRIAL: NCT02140242
Title: Randomized Comparison Between Two Dose Levels of Daunorubicin and Between One Versus Two Cycles of Induction Therapy for Adult Patients With Acute Myeloid Leukemia ≤65 Years
Brief Title: Comparison Between Two Dose Levels of Daunorubicin and Between One vs. Two Induction Cycles for Adult Patients With AML
Acronym: DaunoDouble
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: University Hospital Dresden (Other); Masaryk University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: TUD-2DAUNO-058
Record Dates: First submitted 2014-05-09; First posted 2014-05-16 (Estimated); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Leukemia, Myelocytic, Acute
Keywords: AML; leukemia; induction treatment; daunorubicin; 7+3
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- daunorubicin 60 mg/m2 (Active Comparator): study part 1 - dose daunorubicin standard dose daunorubicin in induction 1 (60 mg/m2) on days 3-5
  Interventions: Drug: study part 1 - dose daunorubicin
- Double induction (Active Comparator): study part 2: induction cycles double induction (only patients with good response)
  Interventions: Procedure: induction cycles
- Single induction (Experimental): study part 2: induction cycles single induction (only patients with good response)
  Interventions: Procedure: induction cycles

INTERVENTIONS:
Drug: study part 1 - dose daunorubicin — standard induction dose of daunorubicin 60 mg/m2 on days 3-5
  Arms: daunorubicin 60 mg/m2
Procedure: induction cycles — single induction cycle versus double induction cycles (only patients with good response after first induction) Allocation is randomized for cytogenetic risk.
  Arms: Double induction; Single induction

SUMMARY:
The proposed trial will address two clinically important questions for younger patients with newly diagnosed acute myeloid leukemia (AML): the optimal dose of daunorubicin in induction therapy and the necessity of a second induction cycle in patients with a good response after the first induction. The primary endpoint is the rate of good responders. Secondary outcomes will be relapse-free survival, overall survival and minimal residual disease kinetics. Patients will be recruited in about 40 treatment centers of the Study Alliance Leukemia study group over a period of 40 months. The results will be of great clinical relevance: First, the study could facilitate the establishment or confirmation of the optimal daunorubicin dose.

DETAILED DESCRIPTION:
In the first part of the trial, patients will be randomly assigned to receive either 90 mg/m2 or 60 mg/m2 daunorubicin in the first induction cycle in addition to standard dosed cytarabine. Assuming a superiority of 90 mg/m2, 436 patients will be recruited. In the second part of the trial, good responders will be randomized to receive either a second or no further induction cycle. Assuming a non-inferiority of the single induction regarding the rate of complete remissions, a number of 360 patients will be included in the second part. Furthermore, in case of a non-inferiority of single versus double induction in good responders, about half of all younger AML patients could be spared a second induction cycle, leading to a reduction in treatment-related mortality, fewer days spent in hospital and improved quality of life.

As a result of the preplanned interim analysis of part I, the sponsor decided to suspend randomization in trial part I and to offer all patients the standard dose of 60 mg/m2 daunorubicin in both induction cycles (part I and II of the trial). Because of this an Amendment was sent to and approved by regulatories and ethics comitee.

The inclusion age was raised to 65 years based on the current German treatment guidelines in which patients up to the age of 65 are considered eligible for intensive induction chemotherapy with DA60 [Onkopedia-Leitlinie 2017].

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed AML other than acute promyelocytic leukemia (APL) according to WHO criteria, i.e. bone marrow aspirate or biopsy must contain ≥20% blasts of all nucleated cells or differential blood count must contain ≥20% blasts. In acute erythroid leukemia, ≥20% blasts in all non-erythroid bone marrow cells. In AML defined by cytogenetic aberrations, the rate of blasts may be <20%. Secondary AMLs are eligible for inclusion.
* Age 18- inkl.65 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Adequate liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:

  * Total bilirubin ≤ 1.5 times the upper limit of normal
  * alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 2.5 times upper limit of normal
  * Creatinine ≤ 1.5 times upper limit of normalExclusion Criteria:
* Adequate cardiac function, i.e. left ventricular ejection fraction (LVEF) of ≥ 50% as assessed by transthoracic two-dimensional echocardiography ("M Mode") or multiple gated acquisition scan (MUGA scan)
* Signed informed consent
* Women must fulfill at least one of the following criteria in order to be eligible for trial inclusion:

  * Post-menopausal (12 months of natural amenorrhea or 6 months of amenorrhea with Serum follicle stimulating hormone (FSH) > 40 U/ml)
  * Postoperative (i.e. 6 weeks) after bilateral ovariectomy with or without hysterectomy
  * Continuous and correct application of a contraception method with a Pearl Index of <1% (e.g. implants, depots, oral contraceptives, intrauterine device - IUD).
  * Sexual abstinence
  * Vasectomy of the sexual partner

Exclusion criteria:

* Patients who are not eligible for standard chemotherapy as assessed by the treating physician
* Central nervous system manifestation of AML
* Cardiac disease: i.e. heart failure New York Heart Association (NYHA) III or IV; unstable coronary artery disease (MI more than 6 months prior to study entry is permitted); serious cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Patients undergoing renal dialysis
* Chronic pulmonary disease with clinical relevant hypoxia
* Known HIV or Hepatitis infection
* Uncontrolled active infection
* Medical conditions other than AML with an estimated life expectancy below 6 months
* Previous treatment of AML except hydroxyurea up to 5 days
* Relapsed or primary refractory AML
* Acute promyelocytic leukemia
* Previous anthracycline-containing chemotherapy
* Treatment with any known non-marketed drug substance or experimental therapy within 4 weeks prior to enrollment
* Incapability of understanding purpose and possible consequences of the trial
* Pregnant or breastfeeding women
* Evidence suggesting that the patient is not likely to follow the study protocol (e.g. lacking compliance)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 721 (Actual)
Dates: Start 2014-04-16 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
response rate after first induction | day 15
  To investigate whether a higher dose of daunorubicin in induction chemotherapy leads to an increase in hematological good responders defined as having <5% myeloid blasts on day 15 after start of induction therapy.
Rate complete remissions | day 35 after final induction
  To investigate whether the rate of complete remissions (CR) after single induction is similar to that after double induction in patients with good response to induction I.

SECONDARY OUTCOMES:
rate cytogenetic and molecular complete remissions | day 35
  To investigate whether a higher dose of daunorubicin in induction chemotherapy will lead to an increase in cytogenetic and molecular complete remissions.
event-free survival (EFS) | 5 years
  To investigate whether a higher dose of daunorubicin will lead to improved event-free survival (EFS), relapse-free survival (RFS) and overall survival (OS). To investigate whether EFS, RFS and OS are similar after single versus double induction in patients with good response to induction I.
relapse-free survival (RFS) | 5 years
  To investigate whether a higher dose of daunorubicin will lead to improved event-free survival (EFS), relapse-free survival (RFS) and overall survival (OS). To investigate whether EFS, RFS and OS are similar after single versus double induction in patients with good response to induction I.
overall survival (OS) | 5 years
  To investigate whether a higher dose of daunorubicin will lead to improved event-free survival (EFS), relapse-free survival (RFS) and overall survival (OS). To investigate whether EFS, RFS and OS are similar after single versus double induction in patients with good response to induction I.
Correlation between Minimal Residual Disease (MRD) and EFS, RFS, OS | day 35
  To correlate the level of cytogenetic and molecular minimal residual disease after induction treatment with survival outcomes EFS, RFS and OS.
Rate of induction deaths | day 60
  Rate of induction deaths (until day 60 or beginning of consolidation treatment - whichever occurs first)
Incidence of serious infectious complications | day 35
  Incidence of serious infectious complications Grades 3-4 (Common Toxicity Criteria for Adverse Effects (CTCAE) V4.0
Sonographic cardiac left ventricular ejection fraction | day 35
  Sonographic cardiac left ventricular ejection fraction
Serum levels of pro-brain natriuretic peptide (por-BNP) and Troponin-T | day 35
  Serum levels of pro-BNP and Trop-T
Incidence of CTCAE grade ≥3 cardiac complications | day 35
  Incidence of CTCAE grade ≥3 cardiac complications
Rate of early deaths | week 2
  Rate of early deaths (2 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Röllig, Prof. Dr., Principal Investigator — Medizinische Fakultät der TU Dresden, Medizinische Klinik und Poliklinik I
Locations (38):
- Czechia (5):
  - Interní klinika LF Masarykovy univerzity a Fakultní nemocnice Brno, Brno
  - Faculty Hospital Hradec Králové, II. Clinic of international medicine, Hradec Králové
  - Fakultní nemocnice Olomouc, Olomouc
  - Fakultní nemocnice Královské Vinohrady, Prague
  - Ústav hematologie a krevní transfuze (ÚHKT), Prague
- Germany (33):
  - Uniklinik RWTH Aachen, Aachen
  - Klinikum Altenburger Land GmbH, Altenburg
  - Klinikum Augsburg, Augsburg
  - Sozialstiftung Bamberg Klinikum am Bruderwald, Bamberg
  - Charite Campus Benjamin Franklin, Berlin
  - Helios Klinikum Berlin-Buch, Berlin
  - Klinikum Bielefeld, Bielefeld
  - Augusta Kliniken Bochum Hattingen, Bochum
  - Ev. Diakonie-Krankenhaus gGmbH Bremen, Bremen
  - Klinikum Chemnitz GmbH, Chemnitz
  - Carl.Thiem-Klinikum Cottbus gGmbH, Cottbus
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Krankenhaus Düren gem. GmbH, Düren
  - Marienhospital Düsseldorf GmbH, Düsseldorf
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Essen, Essen
  - Johann Wolfgang Goethe-Universität Frankfurt am Main, Frankfurt am Main
  - Universitätsklinikum Halle (Saale), Halle
  - Asklepios Klinik St. Georg, Hamburg
  - St. Marien-Hospital Hamm, Hamm
  - Universitätsklinikum Heidelberg, Heidelberg
  - St. Bernward Krankenhaus Hildesheim, Hildesheim
  - Universitätsklinikum Jena, Jena
  - Westpfalz-Klinikum GmbH, Kaiserslautern
  - Städtisches Krankenhaus Kiel, Kiel
  - Gemeinschaftsklinikum Mittelrhein GmbH, Koblenz
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Gießen und Marburg, Marburg
  - Universitätsklinikum Münster, Münster
  - Klinikum Nürnberg-Nord, Nuremberg
  - Diakonie-Klinikum Schwäbisch Hall gGmbH, Schwäbisch Hall
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Rems-Murr-Klinikum Winnenden, Winnenden

REFERENCES:
- [Derived] Dendorfer SM, Schmidt-Brucken K, Kramer M, Steffen B, Schliemann C, Mikesch JH, Alakel N, Herbst R, Hanel M, Hanoun M, Kaufmann M, Weinbergerova B, Schafer-Eckart K, Sauer T, Neubauer A, Burchert A, Baldus CD, Mertova J, Jost E, Niemann D, Novak J, Krause SW, Scholl S, Hochhaus A, Held G, Szotkowski T, Rank A, Schmid C, Fransecky L, Kayser S, Schaich M, Fiebig F, Haake A, Schetelig J, Middeke JM, Stolzel F, Platzbecker U, Thiede C, Muller-Tidow C, Berdel WE, Ehninger G, Mayer J, Serve H, Bornhauser M, Rollig C. Randomized Comparison of Cardiotoxicity With 60 Versus 90 mg Daunorubicin in AML Induction Therapy. Am J Hematol. 2026 Jan 5. doi: 10.1002/ajh.70160. Online ahead of print. PMID 41492073
- See also: study alliance — https://www.aml-germany.com/
- See also: University Hospital — http://www.uniklinikum-dresden.de/
- See also: czech ECRIN center — https://www.czecrin.cz/